CLINICAL TRIAL: NCT07394543
Title: Retrospective French Registry of Cardiovascular Magnetic Resonance Late Gadolinium Enhancement in Patients With Myocarditis
Brief Title: French Registry of CMR Late Gadolinium Enhancement in Myocarditis
Acronym: MYOCARDITI-LGE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251399
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Myocarditis Acute
Keywords: Late Gadolinium Enhancement; Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myocarditis is a major cause of death in young adults and carries substantial morbidity, including a significant risk of progression to dilated cardiomyopathy. Current diagnostic and therapeutic strategies remain poorly defined, making risk stratification crucial to enable personalized treatments and reduce mortality and major cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Ability to provide informed non-opposition
3. AM diagnosis confirmed using CMR, fulfilling the modified Lake Louise diagnostic criteria

Exclusion Criteria:

1. Patients unable to provide informed non-opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all consecutive patients with AM referred for CMR assessment.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2036-02-10 (Estimated); Study Completion 2036-02-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | From enrollment to the end of follow up at 10 years
  All-cause mortality defined using the French national registry of death (INSEE).

SECONDARY OUTCOMES:
All-cause death | From enrollment to the end of follow up at 10 years
Heart transplantation | From enrollment to the end of follow up at 10 years
Ventricular arrhythmia | From enrollment to the end of follow up at 10 years
Hospitalisation for acute heart failure | From enrollment to the end of follow up at 10 years